CLINICAL TRIAL: NCT00258284
Title: Phase II Trial of Capecitabine (Xeloda) and Weekly Docetaxel (Taxotere) in Metastatic Androgen Independent Prostate Carcinoma
Brief Title: Capecitabine and Docetaxel in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ulka Vaishampayan, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000445613; P30CA022453 (NIH); WSU-D-2615; WSU-HIC-067903MP4F
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Cancer
Keywords: recurrent prostate cancer; stage IV prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Capecitabine; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Docetaxel & Capecitabine (Experimental): Patients receive docetaxel IV over 30 minutes on days 1, 8, and 15 and oral capecitabine twice daily on days 5-18. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses of therapy beyond CR
  Interventions: Drug: capecitabine; Drug: docetaxel

INTERVENTIONS:
Drug: capecitabine — Patients receive docetaxel IV over 30 minutes on days 1, 8, and 15 and oral capecitabine twice daily on days 5-18. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses of therapy beyond CR
  Other Names: Xeloda®
Drug: docetaxel — Patients receive docetaxel IV over 30 minutes on days 1, 8, and 15 and oral capecitabine twice daily on days 5-18. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses of therapy beyond CR
  Other Names: Taxotere®

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as capecitabine and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving capecitabine together with docetaxel works in treating patients with metastatic prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate in patients with androgen-independent metastatic adenocarcinoma of the prostate treated with capecitabine and docetaxel.

Secondary

* Determine the toxicity of this regimen in these patients.
* Determine the progression-free survival, time to treatment failure, and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 30 minutes on days 1, 8, and 15 and oral capecitabine twice daily on days 5-18. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients achieving a complete response (CR) receive 2 additional courses of therapy beyond CR

After completion of study treatment, patients are followed periodically for survival.

PROJECTED ACCRUAL: A total of 28 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Metastatic disease
  * Androgen-independent disease
* Progressive disease, as documented by ≥ 1 of the following criteria:

  * Rising prostate-specific antigen (PSA) despite androgen deprivation therapy and anti-androgen withdrawal

    * Demonstrates a rising PSA trend with 2 successive elevations ≥ 1 week apart
  * Measurable disease progression
  * Nonmeasurable disease progression, defined as the following:

    * PSA ≥ 5 ng/mL
    * New areas of bone metastases on bone scan
* Serum testosterone ≤ 0.5 ng/mL (castrate level)

  * Concurrent luteinizing hormone-releasing hormone agonist therapy required for medically castrated patients

PATIENT CHARACTERISTICS:

Performance status

* Zubrod 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count ≥ 1,500/ mm^3
* Hemoglobin ≥ 8.0 g/dL
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin normal
* Transaminases meeting 1 of the following criteria:

  * AST and/or ALT ≤ 2.5 times upper limit of normal (ULN) if alkaline phosphatase (AP) normal
  * AP ≤ 4 times ULN if AST and/or ALT normal

Renal

* Creatinine clearance ≥ 50 mL/min OR
* Creatinine ≤ 2 mg/dL

Cardiovascular

* No congestive heart failure
* No second- or third-degree heart block
* No myocardial infarction within the past 3 months

Other

* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* No other malignancy within the past 2 years except adequately treated skin cancer or other cancer in complete remission
* No history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* No peripheral neuropathy ≥ grade 2

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy for metastatic disease

Endocrine therapy

* See Disease Characteristics
* More than 4 weeks since prior flutamide
* More than 6 weeks since prior bicalutamide or nilutamide

Radiotherapy

* At least 4 weeks since prior radiotherapy

Other

* At least 28 days since prior investigational drugs for prostate cancer
* No other concurrent anti-cancer therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2003-08; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Response rate by RECIST criteria after every 2 courses | at cycle 2 and every other cycle thereafter

SECONDARY OUTCOMES:
Toxicity at 30 days after last treatment | Every week during treatment cycles
Progression-free survival | Every 2 cycles
Time to treatment failure | Every 2 cycles
  From date of registration to date of progressive disease, or date patient is taken off study for any other reason.
Overall survival | Every 2 cycles
Effect of treatment on biological correlates (thymidine phosphorylase, dihydropyrimidine dehydrogenase, thymidylate synthase) | Every week during treatment cycles

CONTACTS AND LOCATIONS:
Overall Officials: Ulka N. Vaishampayan, MD, Study Chair — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States